CLINICAL TRIAL: NCT05525091
Title: Neoneur Feeding System Functionality in the Clinic - Investigating Assessment of Quantifying Feeding Functionality in Premature and Cardiac Surgery Neonates in Comparison to Dr. Medoff-Cooper's Past Research
Brief Title: Neoneur Feeding System Functionality in the Clinic
Acronym: NN200
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neoneur LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NN2022-01; 1R44NR020275-01 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Feeding Patterns; Feeding; Difficult, Newborn; Feeding Disorder Neonatal
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feeding Assessment (Experimental): Feeding assessment of High-risk premature infants
  Interventions: Other: Feeding Evaluation

INTERVENTIONS:
Other: Feeding Evaluation — Feeding Evaluation with Device
  Other Names: Neoneur 200

SUMMARY:
Prospective data collection using the Neoneur Feeding System to demonstrate device functionality, correlation to historic data, and prepare for a more extensive phase II SBIR trial

DETAILED DESCRIPTION:
The consented infant's assigned Speech Language Pathologist will use the Neoneur Feeding System 2-3 times a week from initiation of oral feeding until discharge, if oral feeding is prescribed. It can be used either as a special consult, or during routine care. The feeding is performed by the Speech Language Pathologist assigned to the infant. There will be no change in the infant's feeding plan. For infants consented to participate in the study, their feeding will include the Neoneur feeding system inserted between the nipple and bottle. When the Neoneur is inserted, it will capture both the suck and swallow changes (oral cavity pressure), and respiration (temperature changes) patterns.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants: requiring tube assisted feeding while in the NICU, gestational age at birth =<34 week, extubated by term
* Infants with CHD: requiring surgery during the first month of life, gestational age > 37 weeks

Exclusion Criteria:

* Premature infants: craniofacial anomalies, infants with grade IV intraventricular hemorrhage, apgar < 5 at 5 minutes, short gut syndrome, history of NEC
* Infants with CHD: no other congenital anomalies, no history of major neurologic insult , listed for heart transplant, history of ECMO, intubated for > 4 weeks, requiring additional surgery

Ages: 1 Day to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-08-14 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
Maturation | 6 weeks of data collection
  Neoneur 200 measures are corelated to infant maturation in gestational age
Telehealth functionality | 6 months
  Evaluation of Sending Neoneur 200 data from the bedside to the cloud for used in the hospital and home

SECONDARY OUTCOMES:
Respiratory | 6 months
  The evaluation of Neoneur 200's respiratory sensor to collect accurate data

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Medoff-Cooper, MSN, PhD, Principal Investigator — Children's Hospital of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
the results will be available and we will seek publication